CLINICAL TRIAL: NCT04457739
Title: Evaluation of Tidal Volume Challenge to Detect Preload-responsiveness in Patients With Acute Respiratory Distress Syndrome (ARDS) During Prone Position
Brief Title: Assessment of Preload Responsiveness in ARDS Patients During Prone Position
Acronym: PR-ARDS-PP
Status: Completed | Type: Observational
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Rui Shi, Principal Investigator, Bicetre Hospital
Other Study IDs: 2019-A00064-53
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Distress Syndrome; Septic Shock; Hemodynamic Instability
Keywords: Hemodynamic monitoring; preload responsiveness; ARDS; Fluid therapy
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tidal volume challenge — Increasing tidal volume from 6 to 8 mL/kg during 1 min
Other: End-expiratory occlusion test — Interrupting the ventilator at end-expiration for 15-30 s and assessing the resulting changes in cardiac output
Other: Trendelenburg maneuver — Patients remained in prone position with a 13° upward bed angulation throughout the study and then be positioned in a declining position at -12 ° for 1 minute

SUMMARY:
Evaluation of preload responsiveness in ARDS patients during prone position is difficult and only one study showed Trendelenburg manoeuvre can be used in this group of patients. This study aims to investigate whether end-expiratory occlusion test, tidal volume challenge (using the changes in PPV) can be used to evaluate preload responsiveness in patients with ARDS ventilated with a low tidal volume and who underwent a PP session.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) which is a major cause of morbidity and mortality in the intensive care unit, is characterized by decreased lung volume, decreased lung compliance, increased pulmonary vascular resistance and pulmonary hypertension, which ultimately lead to right ventricular dysfunction. Moreover, through biventricular interdependence and inter-ventricular septum shift, the left ventricular filling is limited, which eventually results in a decrease in stroke volume. Due to the high risk of ventilation-induced lung injury, protective lung ventilation is recommended, mainly through a reduction in tidal volume. However, due to the profound hypoxemia inherent to this mode of ventilation, lung recruitment strategies are recommended. When the application of a recruitive positive end-expiratory pressure fails to correct hypoxemia, prone positioning (PP) is recommended. A randomized controlled trial (PROSEVA) reported that early application of prolonged PP sessions in patients with severe ARDS significantly decreased 28- and 90-day mortality. In addition to its respiratory effects (improvement in arterial oxygenation and lung recruitment), PP exerts different cardiovascular effects. By increasing oxygenation and recruiting lung regions, PP can reduce the right ventricular afterload. By increasing the intraabdominal pressure (IAP), PP can increase the venous return and the cardiac preload. This effect might depend on the level of IAP, because a high IAP might collapse the inferior vena cava, especially in the case of hypovolemia. If cardiac preload increases, the resultant effect on cardiac output might depend on the degree of preload responsiveness. Finally, by increasing the IAP, PP can increase the left ventricular afterload. In a recent clinical study, our group showed that PP increases right and left ventricular preload and decreased right ventricular afterload. However, PP increased cardiac output only in patients with preload responsiveness. In this study preload responsiveness was detected by an increase in cardiac output > 10% during a passive leg raising (PLR) test. Since PP sessions are recommended to last between 16 to 18 hours per day and since patients with ARDS often have an associated sepsis, hemodynamically instability may occur during PP sessions. The therapeutic decision is very tricky since the administration of fluid (the main therapeutic option in case of hemodynamic instability) is risky due to alteration of lung capillary membrane permeability. Thus, it is important to predict the benefits of fluid administration by using indices of preload responsiveness. The recommended indices of preload responsiveness are pulse pressure variation (PPV), stroke volume variation (SVV) and PLR. However, PPV and SVV cannot be used reliably during low tidal volume ventilation. Moreover, conventional PLR cannot be performed during PP. It is thus important to develop other preload responsiveness tests doable during PP. Our group proposed to perform an end-expiratory occlusion (EEO) test to predict fluid responsiveness in the supine position and more recently to perform a tidal volume challenge (TVC) by transiently increasing tidal volume from 6 to 8 mL/kg and observing the changes in PPV.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patient
* Prone position
* Monitored by transpulmonary thermodilution and pulse contour analysis

Exclusion Criteria:

* Age below 18
* No social security
* Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe ARDS (according to the Berlin definition) undergoing a prone position session, already monitored with a transpulmonary thermodilution device and for whom the evaluation of preload responsiveness is needed owing to the occurrence of hemodynamic instability.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Area under ROC curve of the change in pulse pressure variation during tidal volume challenge to detect preload responsiveness | 1 minute after increasing tidal volume from 6 to 8mL/kg

SECONDARY OUTCOMES:
Area under ROC curve of the pulse pressure variation in tidal volume of 8ml/kg in continuous cardiac output during end-expiratory occlusion to detect preload dependence | 1 minute after tidal volume increase to 8 ml/kg

CONTACTS AND LOCATIONS:
Locations (1):
- Bicetre Hospital, Paris, Val-de-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Background] Vieillard-Baron A, Matthay M, Teboul JL, Bein T, Schultz M, Magder S, Marini JJ. Experts' opinion on management of hemodynamics in ARDS patients: focus on the effects of mechanical ventilation. Intensive Care Med. 2016 May;42(5):739-749. doi: 10.1007/s00134-016-4326-3. Epub 2016 Apr 1. PMID 27038480
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Jozwiak M, Monnet X, Teboul JL. Optimizing the circulation in the prone patient. Curr Opin Crit Care. 2016 Jun;22(3):239-45. doi: 10.1097/MCC.0000000000000308. PMID 27101363
- [Background] Jozwiak M, Teboul JL, Anguel N, Persichini R, Silva S, Chemla D, Richard C, Monnet X. Beneficial hemodynamic effects of prone positioning in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1428-33. doi: 10.1164/rccm.201303-0593OC. PMID 24102072
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Guerin C, Beuret P, Constantin JM, Bellani G, Garcia-Olivares P, Roca O, Meertens JH, Maia PA, Becher T, Peterson J, Larsson A, Gurjar M, Hajjej Z, Kovari F, Assiri AH, Mainas E, Hasan MS, Morocho-Tutillo DR, Baboi L, Chretien JM, Francois G, Ayzac L, Chen L, Brochard L, Mercat A; investigators of the APRONET Study Group, the REVA Network, the Reseau recherche de la Societe Francaise d'Anesthesie-Reanimation (SFAR-recherche) and the ESICM Trials Group. A prospective international observational prevalence study on prone positioning of ARDS patients: the APRONET (ARDS Prone Position Network) study. Intensive Care Med. 2018 Jan;44(1):22-37. doi: 10.1007/s00134-017-4996-5. Epub 2017 Dec 7. PMID 29218379
- [Background] Wheeler AP, Bernard GR. Acute lung injury and the acute respiratory distress syndrome: a clinical review. Lancet. 2007 May 5;369(9572):1553-1564. doi: 10.1016/S0140-6736(07)60604-7. PMID 17482987
- [Background] Chiumello D, Brochard L, Marini JJ, Slutsky AS, Mancebo J, Ranieri VM, Thompson BT, Papazian L, Schultz MJ, Amato M, Gattinoni L, Mercat A, Pesenti A, Talmor D, Vincent JL. Respiratory support in patients with acute respiratory distress syndrome: an expert opinion. Crit Care. 2017 Sep 12;21(1):240. doi: 10.1186/s13054-017-1820-0. PMID 28899408
- [Background] Roch A, Guervilly C, Papazian L. Fluid management in acute lung injury and ards. Ann Intensive Care. 2011 May 30;1(1):16. doi: 10.1186/2110-5820-1-16. PMID 21906342
- [Background] Teboul JL, Monnet X, Chemla D, Michard F. Arterial Pulse Pressure Variation with Mechanical Ventilation. Am J Respir Crit Care Med. 2019 Jan 1;199(1):22-31. doi: 10.1164/rccm.201801-0088CI. PMID 30138573
- [Background] Yonis H, Bitker L, Aublanc M, Perinel Ragey S, Riad Z, Lissonde F, Louf-Durier A, Debord S, Gobert F, Tapponnier R, Guerin C, Richard JC. Change in cardiac output during Trendelenburg maneuver is a reliable predictor of fluid responsiveness in patients with acute respiratory distress syndrome in the prone position under protective ventilation. Crit Care. 2017 Dec 5;21(1):295. doi: 10.1186/s13054-017-1881-0. PMID 29208025
- [Background] Sibbald WJ, Paterson NA, Holliday RL, Baskerville J. The Trendelenburg position: hemodynamic effects in hypotensive and normotensive patients. Crit Care Med. 1979 May;7(5):218-24. PMID 467083
- [Background] Geerts BF, van den Bergh L, Stijnen T, Aarts LP, Jansen JR. Comprehensive review: is it better to use the Trendelenburg position or passive leg raising for the initial treatment of hypovolemia? J Clin Anesth. 2012 Dec;24(8):668-74. doi: 10.1016/j.jclinane.2012.06.003. PMID 23228872
- [Background] Myatra SN, Prabu NR, Divatia JV, Monnet X, Kulkarni AP, Teboul JL. The Changes in Pulse Pressure Variation or Stroke Volume Variation After a "Tidal Volume Challenge" Reliably Predict Fluid Responsiveness During Low Tidal Volume Ventilation. Crit Care Med. 2017 Mar;45(3):415-421. doi: 10.1097/CCM.0000000000002183. PMID 27922879
- [Background] Monnet X, Osman D, Ridel C, Lamia B, Richard C, Teboul JL. Predicting volume responsiveness by using the end-expiratory occlusion in mechanically ventilated intensive care unit patients. Crit Care Med. 2009 Mar;37(3):951-6. doi: 10.1097/CCM.0b013e3181968fe1. PMID 19237902
- [Derived] Shi R, Ayed S, Moretto F, Azzolina D, De Vita N, Gavelli F, Carelli S, Pavot A, Lai C, Monnet X, Teboul JL. Tidal volume challenge to predict preload responsiveness in patients with acute respiratory distress syndrome under prone position. Crit Care. 2022 Jul 18;26(1):219. doi: 10.1186/s13054-022-04087-w. PMID 35850771